CLINICAL TRIAL: NCT03453333
Title: 3-dimensional Versus 2-dimensional Laparoscopy Of Ovarian Cyst (LOOC): a Randomized Controlled Trial
Brief Title: 3-dimensional Versus 2-dimensional Laparoscopy of Ovarian Cyst
Acronym: LOOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kangbuk Samsung Hospital (Other)
Responsible Party: Principal Investigator, Taejong Song, Professor, Kangbuk Samsung Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KBSMC 2018-04-023
Record Dates: First submitted 2018-02-27; First posted 2018-03-05 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Laparoscopy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D laparoscope (Experimental): For laparoscopic camera system, a 10-mm ENDOEYE FLEX 3D Deflectable Videoscope (Olympus Corp., Germany) was used in the 3D group.
  Interventions: Procedure: 3D laparoscope
- 2D laparoscope (Experimental): For laparoscopic camera system, a 10-mm 30º IDEAL EYES Laparoscope (Stryker, Kalamazoo, MI, USA) camera was used in the 2D group.
  Interventions: Procedure: 2D laparoscope

INTERVENTIONS:
Procedure: 3D laparoscope — For laparoscopic camera system, a 10-mm ENDOEYE FLEX 3D Deflectable Videoscope (Olympus Corp., Germany) was used in the 3D group.
  Arms: 3D laparoscope
Procedure: 2D laparoscope — For laparoscopic camera system, a 10-mm 30º IDEAL EYES Laparoscope (Stryker, Kalamazoo, MI, USA) camera was used in the 2D group.
  Arms: 2D laparoscope

SUMMARY:
Lack of depth perception and spatial orientation are drawbacks of laparoscopic surgery. The advent of the three-dimensional (3D) camera system enables surgeons to regain binocular vision. The aim of this study was to gain subjective and objective data to determine whether 3D systems are superior to two-dimensional (2D) systems in terms of surgical outcomes.

DETAILED DESCRIPTION:
Elective laparoscopic ovarian cystectomy is established as the treatment of choice for benign ovarian cysts. The advantages of laparoscopic surgery over conventional open surgery are less pain, shorter recovery time, shorter hospital stay, and consequently faster return to normal activity as well as better cosmetic effects. However, laparoscopic surgery is more challenging compared with open surgery, partly because surgeons must operate in a three-dimensional (3D) space through a two-dimensional (2D) projection on a monitor, which results in loss of depth perception and consequently more cognitive workload on the surgeon. In traditional 2D laparoscopic procedures, the surgeon has to mentally transform and process the 2D image into a 3D image using motion parallax through movement of the laparoscope, relative position of instruments, and shading of light and dark. During the past 3 decades, 3D imaging systems have been introduced in and attempt to improve in-depth perception and spatial orientation during minimally invasive surgery. The anticipated advantages for the surgeon are greater accuracy and speed in manual skills, translating to decreased operative time, a reduced learning curve, and enhanced safety.

Nevertheless, studies, to date, examining the potential advantages and disadvantages of 3D versus 2D imaging systems have produced contradictory results. Moreover, there have been no studies exploring the advantage of 3D imaging system in patients undergoing laparoscopic ovarian cystectomy. The aim of this study was to gain subjective and objective data to determine whether 3D imaging systems in the treatment of ovarian cyst are superior to 2D systems in terms of surgical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* age between 19 and 48 years
* American Society of Anesthesiologists physical status (ASAPS) classification I-II
* absence of pregnancy at the time of surgery.

Exclusion Criteria:

* any suspicious finding of malignant ovarian diseases
* any concomitant diseases requiring uterine or upper abdominal surgery
* unavailability of the surgical recording equipment for laparoscopic procedure
* post-menopausal status

Ages: 19 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2018-05-10 (Actual); Primary Completion 2019-03-12 (Actual); Study Completion 2019-03-12 (Actual)

PRIMARY OUTCOMES:
Operative blood loss | At the time of surgery
  Operative blood loss was measured by the anesthesiologists after defining it as the difference between the total amount of suction and irrigation plus the difference between the total gauze weight before and after surgery.

SECONDARY OUTCOMES:
physical demand | At the time of surgery
  The physical demand was evaluated on a scale of 0 to 10 using the question of "How physically demanding was the task?" High score means high physical demand. Low score means low physical demand.
mental demand | At the time of surgery
  The mental demand was evaluated on a scale of 0 to 10 using the question of "How mentally demanding was the task?" High score means high mental demand. Low score means low mental demand.
visually induced motion sickness (VIMS) | At the time of surgery
  The vision-induced motion sickness (VIMS) was assess using the Simulator Sickness Questionnaire (SSQ), in which higher score indicates worse sickness. The maximum and minimum score of SSQ are 48 and 0 points.

CONTACTS AND LOCATIONS:
Overall Officials: Taejong Song, MD PhD, Principal Investigator — Kangbuk Samsung Hospital, Seoul, Republic of Korea
Locations (1):
- Kangbuk Samsung Hospital, Seoul, Jongno-gu, South Korea

IPD SHARING:
Plan to Share IPD: No